CLINICAL TRIAL: NCT04736095
Title: 3 Dimensional Ultrasound in Comparison to Hysteroscopy in Diagnosis of Myomas
Brief Title: 3 Dimensional Ultrasound in Comparison to Hysteroscopy in Myomas
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Other Study IDs: 3D
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D ultrasound for diagnosis of submucous myomas
  Interventions: Diagnostic Test: 3D Ultrasound
- Hysteroscopy for diagnosis of submucous myoma
  Interventions: Diagnostic Test: Hysteroscopy

INTERVENTIONS:
Diagnostic Test: 3D Ultrasound — Doing 3D ultrasound for diagnosis of submucous myoma
  Groups: 3D ultrasound for diagnosis of submucous myomas
Diagnostic Test: Hysteroscopy — Doing hysteroscopy for diagnosis of submucous myoma
  Groups: Hysteroscopy for diagnosis of submucous myoma

SUMMARY:
• three-dimensional saline infusion sonohysterography (3D SIS) was performed in all cases. A sterile Cuscoe speculum was passed, the cervix visualized and cleaned with sterile chlorhexidine solution. A 3.3 mm soft plastic paediatric naso-gastric suction catheter was then passed through the cervix into the uterine cavity without grasping the cervix.

DETAILED DESCRIPTION:
The speculum was removed and a 5 MHz transvaginal 3D ultrasound probe inserted into the vagina (Voluson 730; KretzTechnik, Austria).

ELIGIBILITY:
Inclusion Criteria:

* • Women between 20 and 60 years with abnormal uterine bleeding in form of heavy menstrual bleeding, irregular and heavy menstrual bleeding) diagnosed on non-enhanced two-dimensional ultrasonography with submucous fibroids.

  * Absence of STD, PID, active vaginal bleeding.

Exclusion Criteria:

* Presence of general cause of abnormal uterine bleeding

  * History of drug use that can cause vaginal bleeding (anticoagulants, OCPs, HRT)
  * History of recent hormonal treatment
  * High risk of undergoing hysteroscopy
  * Vaginal, Vulval causes of bleeding

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with submucous myomas
Study Population: Women between 20 and 60 years with abnormal uterine bleeding
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
The accuracy of 3D ultrasound in doiagnosis of submucous myomas in comparison to hysteroscopy | one week
  How many women will be diagnosed by 3D US to have submucous myoma

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (2):
- Egypt (2):
  - Algazeerah, Giza
  - Aljazeera( Al Gazeera) hospital, Giza